CLINICAL TRIAL: NCT01846065
Title: Tobacco Craving and Triggers in Persons With Schizophrenia
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, MPRC, Heidi Wehring, Pharm.D., BCPP, University of Maryland, Baltimore
Other Study IDs: HP-00055208
Record Dates: First submitted 2013-04-02; First posted 2013-05-03 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Smoker; Schizophrenia Diagnosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigators have recently completed a pilot study exploring the safety and efficacy of using a virtual-reality based cue platform to elicit craving in smokers with schizophrenia(SWS)(Wehring et al, unpublished). In this study, participants with schizophrenia (n=16) showed increased attention to cigarettes and changes in craving measures when participating in the VR craving platform. In addition, participants tolerated the VR environment without undue adverse effects or exacerbation of symptoms. Adverse effects from the VR environment did not differ from that in a non-mentally ill population, and included headache, nausea, and dizziness as most commonly occurring factors. Persons in this pilot also showed acceptable rates of Immersion and Presence in the VR environment, showing the potential use of this form of environment for this and other purposes.

In this study, investigators will examine virtual reality cue-reactivity in smokers with schizophrenia, with a focus on the relationship of cue-reactivity with self-identified triggers/cues. Smokers with schizophrenia often identify specific cues that trigger craving. Many of these are environmental (scent, sight of smoking paraphernalia or cigarettes, related objects, or social situations), however, a significant amount of smokers describe emotionally-based factors (sadness, being upset, etc.) as primary cues and triggers. Most methods used to elicit craving in experimental studies are executed via using environmental cues like sight of cigarettes or smoking paraphernalia. It is not known if smokers with schizophrenia(SWS) who are strongly emotionally triggered will be responsive to environmental triggers in a cue-elicited craving platform. This is an important research question, as the testing of anti-craving interventions should be generalizable for use across SWS with differing triggers to smoking. The VR-based environmental program from our pilot study, which includes sight, scent, and social cues, will be used to test pre-identified environmental cues/triggers and their effects on cue-elicited craving in 30 SWS. Subjective reports, mood and emotion measures, and objective physiological measurements will be used to identify and quantify environmental craving responsivity as well as tonic craving.

Given the high prevalence of smoking among individuals with schizophrenia, understanding some of the environmental factors that serve to maintain nicotine dependence is a critical step in improving smoking cessation treatment outcomes. Establishing and validating a model of cue-elicited responsivity will allow future investigations of craving, and ultimately designs for studying the efficacy of anti-craving medications in people with schizophrenia.

ELIGIBILITY:
Inclusion criteria

1. 18-55 year old males and females
2. currently smokes at least 10 cigarettes per day
3. current DSM-IV diagnosis of schizophrenia or schizoaffective disorder and stable medication regimen
4. medically healthy as determined by screening criteria
5. urine cotinine level ≥ 100 ng/ml (NicAlert® reading ≥ 3)
6. agrees to wear a head mounted display (HMD) for up to 45 minutes
7. participant able to complete the Evaluation to Sign Consent (ESC) with a minimum score of 80% on ESC.

Exclusion criteria

1. interest in reducing or quitting tobacco use within the past 3 months
2. treatment for tobacco dependence in the past 3 months
3. use of nicotine replacement products, bupropion, or varenicline in the past 3 months
4. DSM-IV diagnosis of active alcohol or substance abuse in the past 1 month or dependence within the past 6 months
5. current use of any medication that would interfere with the protocol in the opinion of PI or investigators
6. history of head injury, seizures, or stroke
7. pregnant, nursing, or planning to become pregnant during the study
8. positive urine toxicology screen for substances other than those used for therapeutic purposes: Participants who have an initial positive urine toxicology screen for substances other than those used for therapeutic purposes will will have the opportunity to return within two weeks for a second toxicology screen. If at that time the results are again positive, the participant will be excluded

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will include: current smokers with a DSM-IV diagnosis of schizophrenia or schizoaffective disorder. Participants with schizophrenia will be considered on a stable medication regimen if they have received their current antipsychotic medication(s) for at least 6 weeks and the same dose for at least 30 days.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Relationship between pre-identified environmental cues/triggers (social, environmental, or emotional cues) and their effects on the elicitation of craving in smokers with schizophrenia | 1 Week
  Hypothesis: Based on our pilot data, we hypothesize that smokers with schizophrenia who identify specific environmental cues/triggers of smoking will experience greater self-reported craving as reported by craving on a visual analogue scale and a Tobacco Craving Questionnaire scale as well as physiological responsivity (blood pressure, heart rate, skin conductance) when exposed to environmental smoking cues compared to neutral cues, and will differ from the responsivity of smokers who identify primarily emotional cues.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Wehring, Pharm.D., BCPP, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

REFERENCES:
- See also: Maryland Psychiatric Research Center — http://www.mprc.umaryland.edu